CLINICAL TRIAL: NCT00005065
Title: A Phase I Study of Induction Carboplatin / Paclitaxel Chemotherapy, Pre-operative Radiotherapy With Gadolinium Texaphyrin (Gd-Tex), and Surgical Resection in Stage IIIA (N2) Non-small Cell Lung Carcinoma.
Brief Title: Chemotherapy, Radiation Therapy, and Surgery in Treating Patients With Stage IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01401; OSU 0003; OSU-0003; NCI-T99-0073; OSU-99H0355; OSU-T99-0073; CDR0000067669; U01CA076576 (NIH)
Record Dates: First submitted 2000-04-06; First posted 2003-05-07 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Taxes; Carboplatin; motexafin gadolinium; Surgical Procedures, Operative; Congresses as Topic; Radiotherapy; Radiation

ARMS (1):
- Arm I (Experimental): Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours every 3 weeks for 3 courses. Three weeks after completion of induction chemotherapy, patients receive Gd-Tex IV over 30 minutes twice weekly for 10 doses during preoperative radiotherapy. Radiotherapy is administered daily 5 days a week for 5 weeks. Approximately 3.5 weeks after completion of preoperative radiotherapy, patients undergo complete surgical resection. Three hours prior to surgery, patients receive an eleventh dose of Gd-Tex if they do not develop grade 3 or 4 toxicity with the tenth dose. Patients also receive a MRI without contrast prior to surgery. If the tumor is found to be unresectable, patients may receive additional radiation and/or chemotherapy.
  Interventions: Drug: paclitaxel; Drug: carboplatin; Drug: motexafin gadolinium; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
Drug: motexafin gadolinium — Given IV
  Other Names: gadolinium texaphyrin; Gd (III) Texaphryin; Gd-Tex; PCI-0120; Xcytrin
Procedure: conventional surgery — Undergo complete surgical resection
  Other Names: surgery, conventional
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
Phase I trial to study the effectiveness of combining carboplatin and paclitaxel, radiation therapy with gadolinium texaphyrin, and surgery in treating patients who have stage IIIA non-small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as gadolinium texaphyrin may make the tumor cells more sensitive to radiation therapy. Combining chemotherapy, radiation therapy, and surgery may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine and compare the frequency and grade of toxicities with the use of gadolinium texaphyrin as a radiosensitizer at two dose levels during preoperative radiotherapy in patients with stage IIIA non-small cell lung cancer.

II. Measure the tumor, involved lymph nodes, and normal lung concentrations of gadolinium and compare to the image pixel intensity obtained by the 1.5 Tesla MRI in this patient population given this regimen.

OUTLINE: This is a dose escalation study of gadolinium texaphyrin (Gd-Tex).

Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 1-2 hours every 3 weeks for 3 courses. Three weeks after completion of induction chemotherapy, patients receive Gd-Tex IV over 30 minutes twice weekly for 10 doses during preoperative radiotherapy. Radiotherapy is administered daily 5 days a week for 5 weeks. Approximately 3.5 weeks after completion of preoperative radiotherapy, patients undergo complete surgical resection. Three hours prior to surgery, patients receive an eleventh dose of Gd-Tex if they do not develop grade 3 or 4 toxicity with the tenth dose. Patients also receive a MRI without contrast prior to surgery. If the tumor is found to be unresectable, patients may receive additional radiation and/or chemotherapy.

Cohorts of 3-6 patients receive escalating doses of Gd-Tex until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicities.

Patients are followed at 1 month and then every 4 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell carcinoma of the lung
* Surgical staging with mediastinoscopy or anterior thoracotomy required

  * T1-T3, N2, M0
  * Must appear resectable
* Performance status - Karnofsky 70-100%
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal
* Creatinine no greater than 2 mg/dL
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* FEV greater than 0.8 L
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight loss no greater than 10% of total body weight within past 3 months
* No evidence of neuropathy
* No history of allergy to platinum compounds, paclitaxel, porphyrins, or antiemetics appropriate for administration in conjunction with protocol chemotherapy
* No concurrent uncontrolled illness (e.g., active infection)
* No medical contraindication to MRI (e.g., pacemaker or aneurysm clip)
* No G6PD deficiency
* No known history of porphyria
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No prior chest radiotherapy in area of tumor/nodes
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2000-01; Primary Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as that dose at which fewer than one-third of patients experience dose-limiting toxicity (DLT) graded according to CTC version 2.0 | Up to day 119

SECONDARY OUTCOMES:
Concentrations of gadolinium in tumor, tumor involved lymph nodes, normal lung, and blood | Up to day 123
Image pixel intensities in tumor, tumor involved lymph nodes, normal lung, and blood obtained by 1.5 Tesla MRI | Up to day 119

CONTACTS AND LOCATIONS:
Overall Officials: John Grecula, Principal Investigator — Ohio State University
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States